CLINICAL TRIAL: NCT04728984
Title: A Randomized, Double-blind, Placebo-controlled, Multisite Bridging Clinical Study of Nalfurafine Hydrochloride Orally Disintegrating Tablet in the Treatment of Refractory Pruritus in Hemodialysis Patients
Brief Title: A Multi-site Bridging Study of Nalfurafine Hydrochloride Orally Disintegrating Tablet
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSS-Remitch-HD-III-01
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Uremic Pruritus
MeSH Terms: interventions — TRK 820

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nalfurafine Hydrochloride 5μg (Experimental): Oral administration after dinner, once daily for 14 consecutive days
  Interventions: Drug: Nalfurafine Hydrochloride
- Nalfurafine Hydrochloride 2.5μg (Experimental): Oral administration after dinner, once daily for 14 consecutive days
  Interventions: Drug: Nalfurafine Hydrochloride+Placebo
- Placebo (Placebo Comparator): Oral administration after dinner, once daily for 14 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nalfurafine Hydrochloride — Nalfurafine Hydrochloride 2.5μg*2
  ; Oral administration after dinner, once daily for 14 consecutive days
  Arms: Nalfurafine Hydrochloride 5μg
Drug: Nalfurafine Hydrochloride+Placebo — Nalfurafine Hydrochloride 2.5μg+ A placebo pill; Oral administration after dinner, once daily for 14 consecutive days
  Arms: Nalfurafine Hydrochloride 2.5μg
Drug: Placebo — two placebo pills; Oral administration after dinner, once daily for 14 consecutive days
  Arms: Placebo

SUMMARY:
This is a multisite study to evaluate the efficacy, safety and plasma concentration of Nalfurafine Hydrochloride orally disintegrating tablet in the treatment of refractory pruritus in maintenance hemodialysis patients, and to bridge the efficacy data from Japan

DETAILED DESCRIPTION:
This clinical trial is a bridging study. when selecting the subjects, the most appropriate pruritus medication for the subjects was used first.Then, subjects with "existing treatment-resistant" pruritus will continue to receive basic pruritus treatment if the corresponding treatment is not sufficiently effective, and the experimental drug or placebo will be added to this treatment to evaluate the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic renal failure patients who have been on stable dialysis for 3 months or more, receive regular hemodialysis 3 times a week, and expect no significant treatment changes or dramatic changes in their condition during the clinical trial;
2. In the 1 year prior to signing the informed consent, patients who were treated with the following drugs A and/or B: (A) Systematic treatment (oral, injection, etc.) of "prescribed drugs for pruritus" (including antihistamines or antiallergic drugs) for more than 2 weeks consecutively; (B). Use of " prescribed drugs for pruritus" (ointments, etc.) or topical treatment of moisturizers prescribed by physicians;
3. Patients who had received treatment in inclusion criteria (2) but did not respond;
4. When signing the informed consent, the patient is older than 18 years old (including 18 years old), regardless of gender;
5. During the observation period before administration (D8-14), the number of days for which the VAS values were measured at the time of getting up and going to bed should not be less than 5 days, and the average value of the larger VAS values in the morning and evening measurements should not be less than 50 mm;
6. During the observation period before administration (D8-14), The number of days in which the larger VAS value measured in the morning and evening measurements (if there was a missing time in getting up or going to bed, the value which has been measured was selected) is not less than 20 mm, was not less than 5 days;
7. During the observation period before administration (D8-14), the number of days in which the pruritus severity of Hsie-Kawashima's was evaluated at the time of getting up and at the time of going to bed was not less than 5 days, in which the maximum of the pruritus score was not less than 3 (moderate) in the morning and evening measurements was more than half.

Exclusion Criteria:

1. Malignant tumor patients;
2. Patients with mental illness or mental retardation who cannot correctly understand the VAS score and describe their feelings;
3. Patients with alanine aminotransferase (ALT), aspartate aminotransferase (AST) or glutamine transferase (GGT) or total bilirubin higher than twice the upper limit of normal value (ULN) at the screening stage;
4. Patients currently suffering from atopic dermatitis or chronic urticaria;
5. Patients allergic to opioids;
6. Patients with drug or alcohol dependence;
7. Patients who had received light therapy for pruritus within 1 month prior to signing the informed consent;
8. Patients who have participated in a previous clinical study of Nalfurafine Hydrochloride and have taken Nalfurafine Hydrochloride, or who have participated in this clinical study and have been officially enrolled;
9. Participated in other clinical studies (including research drugs and medical devices) within 1 month before signing the informed consent;
10. Pregnant women, lactating women, women who have a positive pregnancy test or who do not agree to use contraception during the study period;
11. Patients who, as determined by the investigator, could not have their VAS score recorded by themselves for any reason;
12. Patients whose comorbidities or previous medical history, as determined by the investigator, would affect the evaluation of this clinical study;
13. After testing, human immunodeficiency virus antibody positive;
14. Other patients judged by the investigator to be unsuitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Variation in VAS of Nalfurafine Hydrochloride versus Placebo | up to 38(+1) days
  The Variation = the mean of the daily maximum VAS value during the observation period before administration(D8-14) - the mean of the daily maximum VAS value during the administration period (D25-31). Only the days on which the VAS values were recorded during the day and night were evaluated.

SECONDARY OUTCOMES:
Variation in pruritus scores based on the Hsie-Kawashima pruritus severity assessment method | up to 38(+1) days
  Pruritus scores were assessed during the observation period before administration(D8-14) and administration period (D25-31), and only the days when pruritus scores were recorded during the day and night were evaluated.
Variation in nocturnal pruritus scores based on the Hsie-Kawashima pruritus severity assessment method (improvement of pruritus-induced sleep disorders). | up to 38(+1) days
  After calculating the mean values of nocturnal pruritus scores during the observation period before administration(D8-14) and administration period (D25-31), the variation was calculated.
Improvement degree of VAS | up to 38(+1) days
  The average VAS value of the observation period before administration (D8-14) and the average VAS value of the administration period (D25-31) were calculated, and the improvement degree was determined as very effective, effective and ineffective according to the variation of the average VAS value.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No